CLINICAL TRIAL: NCT02011087
Title: Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Small Cell Lung Cancer
Brief Title: Bioelectrical Impedance Phase Angle in Predicting Treatment Outcome in Patients With Extensive Stage Small Cell Lung Cancer Receiving First-Line Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00025808; NCI-2013-02339 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99813A (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Extensive Stage Small Cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (bioelectric impedance analysis) (Experimental): Patients undergo bioelectrical impedance phase angle measurement on day 1 of treatment.
  Interventions: Procedure: bioelectric impedance analysis

INTERVENTIONS:
Procedure: bioelectric impedance analysis — Undergo bioelectric impedance analysis
  Other Names: BIA; bioelectric impedance; bioelectric impedance test; bioimpedance analysis

SUMMARY:
This clinical trial studies bioelectrical impedance phase angle in predicting treatment outcome in patients with extensive stage small cell lung cancer receiving first-line chemotherapy. Diagnostic procedures, such as bioelectrical impedance analysis, may help predict a patient's response to treatment for small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the association between phase angle (PA) measurement and progression-free survival (PFS).

SECONDARY OBJECTIVES:

I. To evaluate the association between PA measurement and treatment-related outcomes of treatment response, adverse treatment events, and overall survival (OS).

II. To determine the feasibility of obtaining PA measurements at a single time point in patients undergoing evaluation in thoracic oncology clinics.

OUTLINE:

Patients undergo bioelectrical impedance phase angle measurement on day 1 of treatment.

After completion of study treatment, patients are followed up every 2-3 months for two years.

ELIGIBILITY:
Inclusion Criteria:

* A primary histopathological and/or cytopathological diagnosis of small cell lung cancer (SCLC)
* Diagnosis of extensive stage disease (extensive stage [ES]-SCLC), with stage established by computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET) scan
* Scheduled to receive front-line platinum-based chemotherapy with carboplatin or cisplatin plus etoposide
* Ability to understand and the willingness to sign an institutional review board (IRB)-approved informed consent document

Exclusion Criteria:

* No recent chemotherapy or surgery, as defined as in the last 6 months
* Presence of a pacemaker or defibrillator
* Patients with major chronic disease known to adversely affect PA, including human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS), congestive heart failure, tuberculosis
* Patients with body mass index (BMI) greater than 34 or less than 16
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unable or unwilling to follow protocol requirements
* Pregnant women are excluded from participation due to inability to participate in required chemotherapy regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From the start of treatment to the time of progression, death, or date of last contact, assessed up to 2 years
  Analyzed using Kaplan-Meier plots and a log-rank test to test the difference in progression-free survival and high/low phase angle measures.
Standardized phase angle measure | Baseline
  A Cox proportional hazards model will be used. The standardized phase angle measure will be treated as a continuous measure and baseline characteristics will be included as covariates in the survival model.

SECONDARY OUTCOMES:
Best overall response (complete, partial, progressive disease, stable disease) using the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 2 years
  Logistic regression will be used to analyze the association between standardized phase angle and best overall response.
Overall survival | From the start of treatment to date of death or date of last contact, assessed up to 2 years
  A Cox proportional hazards model will be used.
Incidence of adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 2 years
  For those events that are the most common, the mean standardized phase angle for those experiencing the condition will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Ruiz, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States